CLINICAL TRIAL: NCT01947374
Title: Matrix-encapsulated Arthroscopic Autologous Chondrocyte Implantation Versus Microfractures for Articular Cartilage Regeneration. Randomised Clinical Trial.
Brief Title: Arthroscopic Autologous Chondrocyte Implantation Versus Microfractures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Aldo Izaguirre, Dr./Study Director, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 017-05-INR
Record Dates: First submitted 2012-02-04; First posted 2013-09-20 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Tear; Knee, Cartilage, Articular
Keywords: Cartilage; Articular
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chondrocyte implantation (Experimental): From a previous biopsy, articular cartilage matrix is digested and chondrocytes are cultured in 2 passages until implants with at least 6,000,000 cells are constructed. These constructus of 8 mm in diameter are implanted arthroscopically by means of biodegradable anchor (MINILOK QUICKANCHOR TM from DePuy-Mitek ) located at the defect and tied securely.
  Interventions: Procedure: Matrix encapsulated chondrocyte implantation
- Microfractures (Experimental): Subchondral bone perforations that allow a clot to be formed, and subsequent scar at the cartilage defect area.
  Interventions: Procedure: Microfracture awl

INTERVENTIONS:
Procedure: Matrix encapsulated chondrocyte implantation — Each implant contains 6,000,000 autologous chondrocytes.
  Arms: Chondrocyte implantation
Procedure: Microfracture awl — Is an awl that allow perforation of the subchondral bone.
  Arms: Microfractures

SUMMARY:
This is a phase III, randomised controlled trial of matrix-encapsulated chondrocyte implantation procedure compared to the microfracture procedure in the repair of symptomatic cartilage lesions of the knee. Eligible patients were asked for informed consent preoperatively and randomised for chondrocyte implantation of microfractures. Those patients allocated to the chondrocyte implantation group will be harvested at time of first arthroscopic procedure and concurrent lesions were treated, as meniscus repair, ligament reconstruction, or malalignment corrected. The patients allocated to microfracture will be treated at the time of the only arthroscopic procedure. Both groups will have the same rehabilitation program. Prospective clinical, radiographic and magnetic resonance imaging will be performed as main outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic single chondral lesions of the knee from 1 to 4 cm2.
* Signed patient informed consent.
* Agree to adhere to rehabilitation protocol.

Exclusion Criteria:

* Inflammatory arthritis, septic arthritis, gout, pseudogout, Paget's disease, ochronosis, acromegaly, hemochromatosis, tumors, collagen mutations.
* Total meniscectomy
* Malalignment
* Evidence of osteoarthritis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
MRI T2 Mapping | 24 months
  Special magnetic resonance imaging technique for measurement of collagen and water content, expressed in milliseconds.

SECONDARY OUTCOMES:
Clinical evaluation | 0, 10, 30 days; 3, 6, 9 ,12, 24, 36 months
  Clinical assessment with validated knee scores, and adverse effects register are taken.

CONTACTS AND LOCATIONS:
Overall Officials: Clemente Ibarra, M.D., Principal Investigator — INR; Luis G Ibarra, M.D., Study Chair — INR; Enrique Villalobos, M.D., Study Director — INR; Aldo F Izaguirre, M.D. M.Sc., Study Director — INR
Locations (1):
- National Institute of Rehabilitation, Mexico City, Mexico

REFERENCES:
- [Background] Masri M, Lombardero G, Velasquillo C, Martinez V, Neri R, Villegas H, Ibarra C. Matrix-encapsulation cell-seeding technique to prevent cell detachment during arthroscopic implantation of matrix-induced autologous chondrocytes. Arthroscopy. 2007 Aug;23(8):877-83. doi: 10.1016/j.arthro.2007.05.010. PMID 17681210
- [Background] Ibarra-Ponce de Leon JC, Velasquillo-Martinez MC, Izaguirre A, Villalobos-Cordova E, Masri M, Ibarra-Ibarra LG. [Cartilage repair: cell-based techniques]. Acta Ortop Mex. 2009 Jan-Feb;23(1):38-44. Spanish. PMID 19462773
- [Background] Ibarra C, Izaguirre A, Villalobos E, Masri M, Lombardero G, Martinez V, Velasquillo C, Meza AO, Guevara V, Ibarra LG. Follow-up of a new arthroscopic technique for implantation of matrix-encapsulated autologous chondrocytes in the knee. Arthroscopy. 2014 Jun;30(6):715-23. doi: 10.1016/j.arthro.2014.02.032. Epub 2014 Apr 18. PMID 24746406
- [Derived] Ibarra C, Villalobos E, Madrazo-Ibarra A, Velasquillo C, Martinez-Lopez V, Izaguirre A, Olivos-Meza A, Cortes-Gonzalez S, Perez-Jimenez FJ, Vargas-Ramirez A, Franco-Sanchez G, Ibarra-Ibarra LG, Sierra-Suarez L, Almazan A, Ortega-Sanchez C, Trueba C, Martin FB, Arredondo-Valdes R, Chavez-Arias D. Arthroscopic Matrix-Assisted Autologous Chondrocyte Transplantation Versus Microfracture: A 6-Year Follow-up of a Prospective Randomized Trial. Am J Sports Med. 2021 Jul;49(8):2165-2176. doi: 10.1177/03635465211010487. Epub 2021 May 28. PMID 34048286
- See also: Official site of the INR — http://www.inr.gob.mx